CLINICAL TRIAL: NCT06406933
Title: Saliva Conductivity as A Novel Screening Test for Dry Eye Disease and Sjögren's Syndrome
Brief Title: Salivary Conductivity Screening for Dry Eye Disease and Sjögren's Syndrome
Status: Recruiting | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2022017070
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-05

CONDITIONS: Sjogren's Syndrome; Dry Eye Syndromes
Keywords: dry eye disease; Sjögren syndrome; salivary conductivity; conductivity
MeSH Terms: conditions — Sjogren's Syndrome; Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- new-pSS: Newly diagnosed primary Sjögren's syndrome patients
  Interventions: Drug: Carbomer Gel/Jelly
- Sjögren's syndrome: Patients diagnosed with Sjögren's syndrome and who have undergone treatment: Need to undergo major illness card registration.
  Interventions: Drug: Carbomer Gel/Jelly
- dry eye: Those with symptoms of dry eyes (such as a sensation of foreign bodies in the eyes, sensitivity to light, tearing, etc.) but without symptoms of dry mouth (such as frequent drinking of water).
  Interventions: Drug: Carbomer Gel/Jelly
- normal: Those without symptoms of dry eyes or dry mouth.

INTERVENTIONS:
Drug: Carbomer Gel/Jelly — The drug is for dry eye syndrome by providing temporary relief from discomfort and irritation.
  Groups: Sjögren's syndrome; dry eye; new-pSS

SUMMARY:
Dry eye disease, or keratoconjunctivitis sicca, is one of the most common diseases encountered at ophthalmologic clinics. Patient with dry eye disease commonly presented foreign body sensation, red eye, blurred vision, etc. Numerous treatments for dry eye disease are proposed due to its multifactorial etiology. Sjögren syndrome, which is one of the main etiologies of dry eye disease, is an autoimmune disease characterized by dysfunction of lacrimal and salivary glands. Although dry eye status can be easily examined by ocular surface staining, the methods quantifying salivary flow rate are hard to performed clinically, such as salivary gland scintigraphy and sialometry. Furthermore, disease activity could only rely on serum markers or salivary gland ultrasound. Recently, a portable device measuring salivary conductivity is believed to assess fluid status and renal function. Interestingly, the composition of salivary electrolytes in patients with Sjögren syndrome is different from those with other causes of hyposalivation. Thus, this study aims to evaluate whether salivary conductivity in combination with ocular surface staining can be a non-invasive diagnostic test for primary Sjögren syndrome among people with dry eye disease.

DETAILED DESCRIPTION:
Dry eye disease is prevalent among patients presenting with ocular surface diseases, with rates ranging from 5-50% in recent years. In the United States, approximately sixteen million people are affected by this condition. Dry eye patients often experience ocular surface damage, such as punctate epithelial keratitis, superior limbic keratoconjunctivitis, and filamentary keratitis, due to impaired tear lubrication of the cornea. The etiology of dry eye disease is multifactorial, making diagnosis challenging and requiring comprehensive medical history inquiry and various ocular surface staining techniques. In Taiwan, fluorescein strips are commonly used to assess corneal damage severity and tear break-up time to evaluate tear film abnormalities. Recent research utilizing in vivo confocal microscopy has revealed lower sub-basal nerve fiber numbers and higher dendritic cell densities in the cornea of dry eye patients with immune causes.

Dry eye disease was redefined as a multifactorial condition at the International Dry Eye Workshop II (DEWS II) in 2017, categorized into aqueous deficient dry eye (ADDE) and evaporative dry eye (EDE). In Taiwan, Sjögren's Syndrome (SS) is a primary cause of aqueous deficient dry eye, occurring in approximately 4.8% of dry eye disease patients. SS is a chronic autoimmune disease characterized by lymphocyte infiltration of exocrine glands like the salivary and lacrimal glands. If SS occurs without other autoimmune diseases, it is referred to as primary Sjögren's Syndrome (pSS). Globally, the prevalence of pSS is approximately 60.82 per 100,000 people, with an incidence rate of 6.92 per 100,000 people. Conventional diagnostic methods for salivary dysfunction, such as salivary scintigraphy and parotid sialography, are costly and time-consuming. Following SS diagnosis, comprehensive blood tests, including CBC, DC, ESR, CRP, BUN, Cre, Na, K, HCO3, and serum immunomarkers (ANA, anti-SSA/Ro, anti-SSB/La, RF), are typically advised. The study aims to investigate saliva conductivity as a diagnostic and disease activity monitoring tool for primary Sjögren's syndrome in dry eye syndrome patients and its association with ocular surface damage and tear secretion volume.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 20 and older
2. Patients with normal and dry eye syndrome

Exclusion Criteria:

1. Hepatitis C
2. Acquired immunodeficiency syndrome
3. Lymphoma
4. Intestinal amyloidosis
5. Open pulmonary tuberculosis
6. Graft-versus-host disease
7. Rheumatoid or lupus erythematosus and other autoimmune diseases
8. IgG4-related diseases
9. Head and neck radiation therapy
10. Glaucoma
11. History of infectious keratitis
12. History of ophthalmic surgery
13. Wear contact lenses in the month before the trial
14. Chew betel nuts or smoke within one month before the trial

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We recruited adults aged 20 years and older from the outpatient department and divided them into groups.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Ocular Surface Disease Index (OSDI) questionnaire | 2023-2025
  To evaluate the severity of dry eye symptoms.Thus, the OSDI is scored on a scale of 0 to 100, with higher scores representing greater disability.

SECONDARY OUTCOMES:
Tear Film Break-up Time | 2023-2025
  to indicate the stability of tear film

OTHER OUTCOMES:
Schirmer test | 2023-2025
  to assess tear production.

CONTACTS AND LOCATIONS:
Overall Officials: PeiLun Wu, Principal Investigator — Chang Gung Memorial Hospital; YungKang Chen, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Department of Ophthalmology, Chang Gung Memorial Hospital, Pizi, Taiwan